CLINICAL TRIAL: NCT02962505
Title: Continuous Regional Analysis Device for Neonate Lung
Acronym: CRADL
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Middlesex University London (Unknown); University College, London (Other); NICU of Makarios III Hospital-The Ministry of Health for the Republic of Cyprus (Unknown); Bio-Medical Research Foundation (Unknown); University of Geneva (Unknown); Linneuniversitetet (Unknown); SWISSTOM AG (Unknown); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Studio Fifield (Unknown); Panaxea (Other)
Responsible Party: Principal Investigator, Inez Frerichs, Prof. Dr. Inéz Frerichs, University Hospital Schleswig-Holstein
Other Study IDs: 668259
Record Dates: First submitted 2016-11-03; First posted 2016-11-11 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Infant Respiratory Distress Syndrome; Acute Bronchiolitis; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to assess whether Electrical Impedance Tomography (EIT) has the potential to optimize the ventilator therapy, validate the effectiveness, efficacy and safety of nursing and medical interventions (endotracheal suctioning, posture changes, surfactant therapy, recruitment manoeuvres, etc.) and for early recognition of complications like pneumothorax and endotracheal tube misplacement. The study design is purely observational.

DETAILED DESCRIPTION:
EIT data will be recorded during 72 hours of routine clinical treatment. To prevent any decisions based on EIT information, the clinicians will be blinded to the EIT findings during the study period. Data on clinical interventions and clinical findings will be recorded using a specially adapted graphical user interface on the EIT device in combination with a paper-based case report form (CRF). EIT data analysis will be performed off-line.

ELIGIBILITY:
Inclusion Criteria:

* Written, informed consent of both parents or legal representative
* Admission in the NICU or PICU
* Patients with or at high risk of developing respiratory failure needing respiratory support.

  o i.e. (oxygen need (FiO2>25%) AND noninvasive or invasive respiratory support) AND/OR repeated apnea with desaturations
* Age from birth to 7 years o Initial focus will be on neonates up to 6 kg and 12 months age. Infants of higher weight up to 7 years age will be included as EIT belts for this age group become available.

Exclusion Criteria:

* Post menstrual age less than 25 weeks
* Body weight < 600 g
* Electrically active implants
* Thorax skin lesions
* Prior participation for the same diagnosis of lung disease

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study specifically focuses on the EIT monitoring of preterm and term neonates, small infants and children up to the age of 7 years treated in NICU and PICU as this is the population where the need for regional lung function monitoring tools is most urgently needed to optimize the ventilator therapy, validate the effectiveness, efficacy and safety of nursing and medical interventions (endotracheal suctioning, posture changes, surfactant therapy, alveolar recruitment, etc.) and prevent/minimize the occurrence of acute (pneumothorax, endotracheal tube misplacement) and chronic (chronic lung disease or bronchopulmonary dysplasia) adverse effects.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-11; Primary Completion 2019-03-03 (Actual); Study Completion 2019-03-03 (Actual)

PRIMARY OUTCOMES:
Change in aggregate measure of ventilation homogeneity (coefficient of variation and global inhomogeneity index of regional tidal volume) by > 10% compared with baseline | 72 hours
Change in right-to-left and/or anteroposterior ventilation distribution by >10% compared with baseline | 72 hours
Time and duration of right-to-left or left-to-right ventilation ratio >2:1 | 72 hours
Percentage of EIT examination time with at least 26 out of 32 sensors exhibiting skin contact impedance of < 700 Ohm | 72 hours
  Skin contact impedance will be monitored continuously by the EIT device. If more than 6 sensors exhibit skin contact impedance > 700 Ohm, the examination is no longer suitable for analyzing. To assess the percentage of EIT measurements suitable for analyzing, we will calculate the percentage of EIT examination time with at least 26 out of 32 sensors exhibiting skin contact impedance of less than 700 Ohm.

SECONDARY OUTCOMES:
Relationship between time of onset/end of non-invasive respiratory support and EIT findings | 72 hours
Relationship between time of intubation/extubation and EIT findings | 72 hours
Relationship between time of suctioning and EIT findings | 72 hours
Relationship between time and type of posture change and EIT findings | 72 hours
Relationship between time of surfactant administration and EIT findings | 72 hours
Relationship between time of clinically indicated radiological examination and EIT findings | 72 hours
Relationship between time of recruitment manoeuvre and EIT findings | 72 hours
Relationship between time of confirmed pneumothorax and EIT findings | 72 hours
Relationship between time of confirmed endotracheal tube malposition and EIT findings | 72 hours
Relationship between primary cause of respiratory failure and EIT findings | 72 hours
Relationship between fraction of inspired oxygen over time and EIT findings | 72 hours
Relationship between saturation of peripheral oxygen over time and EIT findings | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Inez Frerichs, MD, Study Chair — University Medical Center SH, Kiel , Germany
Locations (4):
- Archbishop Makarios III Hospital, Nicosia, Cyprus
- Oulu University Hospital, Oulu, Finland
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - VU University Medical Center, Amsterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Becher TH, Miedema M, Kallio M, Papadouri T, Karaoli C, Sophocleous L, Rahtu M, van Leuteren RW, Waldmann AD, Strodthoff C, Yerworth R, Dupre A, Benissa MR, Nordebo S, Khodadad D, Bayford R, Vliegenthart R, Rimensberger PC, van Kaam AH, Frerichs I. Prolonged Continuous Monitoring of Regional Lung Function in Infants with Respiratory Failure. Ann Am Thorac Soc. 2022 Jun;19(6):991-999. doi: 10.1513/AnnalsATS.202005-562OC. PMID 34898392